CLINICAL TRIAL: NCT03732573
Title: Can Brief Text Messages Based on Control Theory Promote the Use of Bike Share Schemes?
Brief Title: Can Brief Text Messages Promote Cycling?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Onur Cem Dogru, Principle Investigator, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: University of Sheffield
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Sedentary Lifestyle
Keywords: Physical Activity; Cycling; Behaviour Change Techniques
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: After completing an online questionnaire, participants will be randomized to intervention or control condition. Participants in the intervention condition will receive text messages designed to promote goal setting in the first week, text messages designed to promote goal operating in the second week, and message designed to promote self-monitoring messages in the third week. All text messages will seek to encourage usage of shared bike schemes (e.g. "How many times can you use a shared bike scheme over the next week? Set yourself a goal and challenge yourself!"). Control group participants will receive no messages during the course of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will receive 9 text messages over 3 weeks. Messages will be based on goal-setting in the first week, goal-operating in the second week, and self-monitoring in the third week.
  Interventions: Behavioral: Text messages
- Control Group (No Intervention): Participants in this group will receive no messages during the intervention period.

INTERVENTIONS:
Behavioral: Text messages — Text messages conveying 3 specific behaviour change techniques
  Arms: Intervention Group

SUMMARY:
Cycling behaviour is not widely adopted despite the known benefits for individuals (e.g. health), communities (e.g. less traffic), and environment (e.g. less pollution). Promoting cycling has been studied with infrastructural changes such as building new paths, segregating cycling and vehicle traffic, placing more traffic signs, etc. Few studies using psychological aspects to promote physical activity indicate that goal setting, goal operating, and self-monitoring techniques to be the most effective ones. Current study aims to convey these techniques via short text messages in order to promote bike share schemes.

DETAILED DESCRIPTION:
BCTs have been used to promote many different behaviours including physical activity. Reviews show that the most effective techniques for promoting physical activity are self-monitoring, intention formation, feedback on performance, and goal setting. These techniques are also the core tenets of control theory, which suggests that setting, monitoring, and operating on goals are central to self-control.

To date, most of the intervention studies targeting psychological predictors of behaviour have used one-to-one communication by professionals, counselling, incentives etc. However, such methods may be difficult and costly to implement on a large scale. The proposed research therefore tests whether delivering these techniques via a convenient method (i.e. SMS text messages) is effective in promoting use of bike share schemes. We will also test whether the strength of participants' intentions to use bike share schemes moderates the effects of the intervention.

Participants will be randomly allocated into one of two groups (one experimental and control group). Participants in the control group will receive no messages. Participants in the intervention group will receive text messages prompting goal-setting (e.g. "How many times can you use a shared bike scheme over the next week? Set yourself a goal and challenge yourself!"), goal operating (e.g. "Make plans about when you could use a shared bike scheme, such as at a particular time or for a particular journey next week."), and self-monitoring (e.g. "Studies show that keeping track of progress can help people to achieve their goals. This is what the apps provided by the shared bike schemes can do for you!"). The messages will comprise of 160 characters at most and participants in the intervention group will receive three messages per week.

One month after taking the baseline survey, participants will be asked to fill in a follow-up survey which will ask them how many times they have used bike share schemes in total during the past month. This information is provided in the apps in "My Trips" section and participants will be asked to count the number of individual trips that they have taken since they completed the baseline survey. It is hypothesized that participants in the intervention group will use bike share schemes more frequently than those in the control group and that the intervention effect will be moderated by the strength of participants' initial intentions.

Mixed-measures (condition x time) ANOVA will be used to test for differences in shared bike use between the groups between baseline and follow-up. A moderation analysis will also be conducted to test whether the effect of the text messages on bike scheme use differs by intention strength.

ELIGIBILITY:
Inclusion Criteria:

* Adults who live in a city with a bike share
* Owns a smart phone

Exclusion Criteria:

* Individuals who cannot ride a bicycle

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in total number of times bike share schemes used before and after the intervention | One month
  Participants will be asked to count number of times they used bike share schemes, which are recorded by phone apps automatically. This will be asked at baseline and follow up questionnaires one month apart.

SECONDARY OUTCOMES:
Use of bike schemes in the past seven days | One week
  Participants will be asked to count number of times they used bike share schemes over the last week (will be asked in the follow up questionnaire which will be send 1 month after the baseline questionnaire). As our intervention takes three weeks and our follow up will be at the end of the month, we wanted to specify use of bike share schemes in the last week without any messages sent.
Change in total number of times participants used their own bike in the past month | One month
  Participants will be asked how many times they used their own bikes in the past month. We want to measure how our intervention affects use of personal bikes. This will be compared with baseline scores for those who reports owning a bicycle.
Use of one's own bike in the past seven days | One week
  Participants will be asked how many times they used their personal bicycles in the past seven days. Similar to use of bike share schemes in the past week, we also want to control for personal bike use in the past week (after all our messages will be sent).

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized dataset could be made available to other researchers.

REFERENCES:
- [Background] Carver CS, Scheier MF. Control theory: a useful conceptual framework for personality-social, clinical, and health psychology. Psychol Bull. 1982 Jul;92(1):111-35. No abstract available. PMID 7134324
- [Background] Bird EL, Baker G, Mutrie N, Ogilvie D, Sahlqvist S, Powell J. Behavior change techniques used to promote walking and cycling: a systematic review. Health Psychol. 2013 Aug;32(8):829-38. doi: 10.1037/a0032078. Epub 2013 Mar 11. PMID 23477577
- [Background] Michie S, Abraham C, Whittington C, McAteer J, Gupta S. Effective techniques in healthy eating and physical activity interventions: a meta-regression. Health Psychol. 2009 Nov;28(6):690-701. doi: 10.1037/a0016136. PMID 19916637
- [Background] Rose T, Barker M, Maria Jacob C, Morrison L, Lawrence W, Strommer S, Vogel C, Woods-Townsend K, Farrell D, Inskip H, Baird J. A Systematic Review of Digital Interventions for Improving the Diet and Physical Activity Behaviors of Adolescents. J Adolesc Health. 2017 Dec;61(6):669-677. doi: 10.1016/j.jadohealth.2017.05.024. Epub 2017 Aug 16. PMID 28822682
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568